CLINICAL TRIAL: NCT03939676
Title: Evaluating Motivation and Reward Mechanisms and Brain Substrates in Adults With Obesity: Further Evidence That Obesity Affects Physical and Mental Health
Brief Title: Evaluating Motivation and Reward Mechanisms and Brain Substrates in Adults With Obesity
Status: Completed | Type: Observational
Sponsor: Brain and Cognition Discovery Foundation (Other)
Responsible Party: Principal Investigator, Roger McIntyre, Executive Director, Brain and Cognition Discovery Foundation
Other Study IDs: Pro00032575
Record Dates: First submitted 2019-04-25; First posted 2019-05-07 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Anhedonia; Obesity
MeSH Terms: conditions — Anhedonia; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major Depressive Disorder or Bipolar Disorder: All eligible participants will be included in this single study arm.

SUMMARY:
Anhedonia and abnormalities in reward behavior are core features of overweight/obesity (OW), a highly prevalent condition within MDD populations, and is independently associated with reward disturbances. The investigators therefore aim to investigate the brain substrates subserving reward and motivation in adults with overweight/obesity.

The primary aim of this pilot study is to determine whether associations exist between obesity and decreased performance on the respective motivation/reward paradigms.

DETAILED DESCRIPTION:
Herein, the investigators are primarily interested in three overlapping, yet distinct aspects, of anhedonia. The investigators are primarily interested in motivation, reward valuation, and reward learning towards addressing the measurement of each of these respective subdomains, eligible participants will complete validated gold standard measures (i.e. the Effort Expenditure for Rewards Task (EEfRT) (reward valuation), Probabilistic Reward Task (PRT) (reward learning), and the Monetary Incentive Delay (MID) task (reward anticipation)).

Twenty adults with overweight/obesity will complete all tasks at a single visit with two of the tasks being completed prior to MRI and one of the tasks (i.e. EEfRT) will be completed during MRI acquisition.

The primary aim of this pilot study is to determine whether associations exist between obesity and decreased performance on the respective motivation/reward paradigms. In addition, associations between performance on reward tasks and functional connectivity, as measured by MRI and DTI, a secondary objective is to ascertain whether associations exist between performance on the motivation reward tasks and gold standard measures of food intake (i.e. food diary) and energy expenditure (i.e. calorimetry).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Meeting DSM-V criteria for: (i) Major depressive disorder (symptomatic or asymptomatic in any phase of the illness) or (ii) bipolar disorder I/II (symptomatic or asymptomatic in any phase of the illness)
* Ability to provide written and informed consent
* Obesity 30 kg/m2
* Weight under 440lbs
* Shoulder-to-shoulder width under 60 cm

Exclusion Criteria:

* Age below 18 or above 65
* Use of benzodiazepines or consumption of alcohol within 12 hours of assessments
* Abuse of marijuana
* Physical, cognitive, or language impairments sufficient to adversely affect data derived from assessments
* Diagnosed reading disability or dyslexia
* Clinically significant learning disorder by history
* History of moderate or severe traumatic brain injury
* Other neurological disorders, or unstable systemic medical diseases
* Pregnancy and post-partum period
* Presence of any contra-indications for MRI
* Weight above 440lbs
* Shoulder-to-shoulder width greater than 60 cm.

All subjects will be consented prior to initiating the study; >45 BMI; suicidality as determined by clinical discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified at the Brain and Cognition Discovery Foundation (BCDF). Twenty subjects between the ages of 18-65 years with obesity, will be enrolled. All patients will be assessed for concurrent psychiatric disorders (e.g. mood disorders) and will meet DSM-V criteria for either: major depressive disorder (symptomatic or asymptomatic in any phase of the illness) or bipolar disorder I/II (symptomatic or asymptomatic in any phase of the illness).
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Effort Expenditure for Rewards Task (EEfRT) | 1 day
  The EEfRT task is a behavioural paradigm that is used to investigate the subject's effort-based decision-making. Subjects are presented with a series of repeated trials wherein they must choose between performing a hard task or an easy task in order to receive monetary compensation (subject's will receive greater compensation for completing the hard task and less compensation for completing the easy task). By presenting the subject with different probability levels for reward receipt, the objective is to examine the extent to which the relationship between motivation (i.e., anhedonia) and effort-based decision-making is modulated by perceived reward magnitude.
Monetary Incentive Delay (MID) Task | 1 day
  The MID is a behavioural paradigm that assesses the basis of anticipation and consumption of reward and punishment. Each run of the MID task consists of approximately 72 trials. The types of cues presented include: circles (indicating the potential to win money i.e., gain cue), squares (indicating the potential to lose money i.e., loss cue), and a triangle (indicating no money will be won or lost i.e., neutral cue). A cue is presented for 500 ms, followed by a fixation cross (2,000 to 2,500 ms) and then the target square (160 to 260 ms), during which the participant is instructed to press a button as quickly as possible to win or avoid losing money. A feedback screen (1,650 ms), in which the top number indicates the amount of money won or lost during that trial, and the bottom number indicates the participant's total amount, is presented at the end of each trial.
Probablistic Reward Task (PRT) | 1 day
  The PRT is a behavioural paradigm that measures response bias and sensitivity to reward under variable conditions. In this task, a signal detection approach is used, whereby subjects must discriminate between two non-ambiguous stimuli displayed rapidly on a computer screen in order to receive a monetary reward. Unbeknownst to the subjects, correct identification of one stimulus is reinforced three times more frequently than the other stimulus. Under these experimental circumstances, healthy subjects reliably develop a response bias for the stimulus that is reinforced more frequently, regardless of which stimulus was actually presented. Thus, reward responsiveness assessed in this task reflects the rapid shaping of future behavioral choices based on prior reinforcement experiences.

SECONDARY OUTCOMES:
MRI/DTI | 1 day
  The secondary outcome will be the association between the EEfRT and function reciprocity of the reward circuit/cognitive control network as measured by MRI/DTI.
  Subjects will be scanned using a 3.0-Tesla Signa HDx scanner with an 8-channel phased-array receiver coil consisting of a structural and functional neuroimaging, comprising:
  1. Whole-brain 3-D T1-weighted Inversion-Recovery prepared Fast Spoiled Gradient-Echo anatomical scan
  2. Whole-brain, T2*-weighted BOLD echo planar imaging during awake resting state
  3. Three runs of whole-brain, T2*-weighted BOLD EPI series during task-based reward paradigm.
  Graph theoretical analysis will be used to assess functional connectivity of the default mode network, cognitive control network, affect network and reward network.
  Associations between obesity and alterations in functional connectivity will be the outcome of interest.

CONTACTS AND LOCATIONS:
Locations (1):
- Canadian Rapid Treatment Centre of Excellence, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03939676/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT03939676/ICF_001.pdf